CLINICAL TRIAL: NCT01676818
Title: Phase II Clinical Trial of Eribulin in Advanced or Recurrent Cervical Cancer
Brief Title: Eribulin Mesylate in Treating Patients With Advanced or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5C-11-2; NCI-2012-01378 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Cervical Cancer; Stage IIIA Cervical Cancer; Stage IIIB Cervical Cancer; Stage IVA Cervical Cancer; Stage IVB Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eribulin mesylate (Experimental): Eribulin mesylate 1.4 mg/m2 IV bolus over 2-5 minutes on days 1 and 8 every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: eribulin mesylate

INTERVENTIONS:
Drug: eribulin mesylate — Given IV
  Other Names: B1939; E7389; ER-086526; halichrondrin B analog

SUMMARY:
This phase II trial studies how well eribulin mesylate works in treating patients with advanced or recurrent cervical cancer. Drugs used in chemotherapy, such as eribulin mesylate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the activity of eribulin (eribulin mesylate) in the management of advanced or recurrent cervical cancer (progression-free survival [PFS].

SECONDARY OBJECTIVES:

I. To describe the toxicity profile of eribulin in patients with advanced or recurrent cervical cancer.

II. To estimate the survival of patients with advanced or recurrent cervical cancer treated with eribulin.

III. To evaluate potential correlative studies as predictive or prognostic makers in this patient population (glucose-regulated protein 78 [GRP78] levels in tissue and blood, tumor protein p53 [p53] expression, apoptosis with terminal deoxynucleotidyl transferase dUTP nick end labeling [TUNEL] assay, apoptosis-related proteins B-cell lymphoma 2 [Bcl-2] and Bcl2-associated X protein [Bax] using immunohistochemistry [IHC], proliferation with Ki-67 IHC, and expression levels of microtubule-associated variables, including tau protein, total alpha- and beta-tubulin, and classes II-IV beta-tubulin isotopes with IHC.

OUTLINE: Patients receive eribulin mesylate 1.4 mg/m2 intravenously (IV) bolus over 2-5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of invasive cervical cancer
* Measurable disease
* 0-1 prior chemotherapy regimens for recurrent or advanced disease; platinum based chemotherapy administered as a radiation sensitizer agent is allowed and does not count as prior therapy
* Absolute granulocyte count (AGC) >= 1,500
* Platelet >= 100,000
* Serum creatinine < 2.0 mg/dl
* Bilirubin =< 1.5 times the upper limit of the normal range (ULN)
* Alkaline phosphatase =< 3 x ULN (in the case of liver metastases, =< 5 x ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (in the case of liver metastases, =< 5 x ULN)
* Peripheral neuropathy grade 0-2
* Recovery of all chemotherapy or radiation-related toxicities to grade =< 1, except for alopecia and peripheral neuropathy
* Performance status 0-2
* Signed informed consent

Exclusion Criteria:

* Prior treatment with eribulin
* Chemotherapy, radiation, or biological or targeted therapy within 3 weeks
* Hormonal therapy within 1 week
* Any investigational drug within 4 weeks
* Known brain metastases, unless previously treated and asymptomatic for 3 months and not progressive in size or number for 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-08-09 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Roman, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was opened to accrual in August 2012 and closed in April 2018. All patients were seen and treated at USC Norris Comprehensive Cancer Center and/or at Los Angeles County + University of Southern California Medical Center.
Pre-assignment Details: The study has no pre-assignment criteria.
Period: Overall Study
Arm/Group | Eribulin Mesylate
Started | 32
Completed | 30
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 32
Disease Type [Count of Participants; unit: Participants] — The number of patients for each disease type was collected and reported in the below sections.
  Participants
    Adenocarcinoma | 8
    Adenosquamous Carcinoma | 1
    Small Cell Carcinoma | 1
    Squamous Cell Carcinoma | 22
Disease Status [Count of Participants; unit: Participants]
  Recurrent | 21
  Advanced | 11
Patient Received Prior Chemotherapy [Count of Participants; unit: Participants] — Per inclusion criteria, patients may have up to 1 prior chemotherapy regimen for recurrent or advanced disease prior to beginning this study.
  Yes = patient received a prior chemotherapy; No = patient did not receive prior chemotherapy.
  Participants
    Yes | 29
    No | 3
Received Prior Regimens [Count of Participants; unit: Participants]
  Cisplatin + Paclitaxel + Bevacizumab | 12
  Cisplatin + Gemcitabine | 12
  Carboplatin + Paclitaxel | 2
  Cisplatin with/without Premetrexed or Capecitabine only | 3
  No Prior Regimen | 3
Received Prior Paclitaxel (PTX) [Count of Participants; unit: Participants]
  Yes | 14
  No | 18
Received Prior Radiation Therapy [Count of Participants; unit: Participants]
  Yes | 28
  No | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival measures the length of time a patient with cancer does not experience disease progression or death. It is defined as the time from first day of treatment to the first observation of disease progression or death due to any cause. If a patient has not progressed or died, progression-free survival is censored at the time of last follow-up.
Time Frame: From the first day of treatment to the first observation of disease progression or death due to any cause, assessed at 6 months
Population: All participants are included
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 32
Months | 2.5 [1.2 to 4.2]

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Safety evaluation according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.3 was used to grade all SAEs. Grade 3+ hematologic and non-hematologic toxicities are reported.
Time Frame: At study drug administration until 30 days following the last dose. Assessed up to 2 years.
Population: All patients who were enrolled and treated with at least 1 dose of the study drug were assessed for safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 32
Participants | 25

3. Secondary Outcome: Best Overall Response (BOR)
Description: BOR is defined as the best response recorded from the start of treatment until disease progression/recurrence, evaluated according to Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1 for target lesions and assessed by MRI: Complete Response (CR) = Disappearance of all target lesions; Partial Response (PR) = at least a 30% decrease in the sum of the diameters of the target lesions compared to the baseline; Stable Disease = Neither enough shrinkage for PR nor enough growth for PD; Progressive Disease = at least a 20% increase in the sum of the diameters of the target lesions from the smallest measurement recorded, with an absolute increase of at least 5 mm, or the appearance of one or more new lesions.
Time Frame: Every 6 weeks from start of treatment until occurrence of progressive disease, assessed up to 4 years.
Population: All patients who received at least 1 cycle of treatment are included. 2 patients were excluded due to not being evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 30
Participants
  Complete Response | 1
  Partial Response | 5
  Stable Disease | 13
  Progressive Disease | 11

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from first day of treatment to time of death due to any cause. If a patient is still alive, survival time is censored at the time of last follow-up.
Time Frame: From first day of treatment to time of death due to any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 32
Months | 6.5 [4.5 to 12.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject received the initial study drug administration and continued until 30 days after the last dose or until resolution of adverse event if beyond 30 days after last dose. Assessed up to 2 years.
Arm/Group | Eribulin Mesylate
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 25/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=32)
Abdominal Pain (Gastrointestinal disorders) | 3
Anemia (Blood and lymphatic system disorders) | 14
Anorexia (Metabolism and nutrition disorders) | 1
Aspartate Aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Hematuria (Renal and urinary disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Paresthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 2
Seizure (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 2
Sinus tachycardia (Cardiac disorders) | 1
Skin infection (Infections and infestations) | 1
Thromboembolic event (Vascular disorders) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Urinary tract obstruction (Renal and urinary disorders) | 1
Urostomy obstruction (Injury, poisoning and procedural complications) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
White blood cell decreased (Investigations) | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=32)
Abdominal Pain (Gastrointestinal disorders) | 16
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 13
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 27
Anal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 29
Anorexia (Metabolism and nutrition disorders) | 26
Anxiety (Psychiatric disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Aspartate Aminotransferase increased (Investigations) | 7
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 20
Bloating (Gastrointestinal disorders) | 1
Blurred vision (Eye disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 9
Bruising (Injury, poisoning and procedural complications) | 4
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Burn (Injury, poisoning and procedural complications) | 1
Chills (General disorders) | 13
Constipation (Gastrointestinal disorders) | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Creatinine increased (Investigations) | 5
Cystitis noninfective (Renal and urinary disorders) | 7
Depression (Psychiatric disorders) | 5
Diarrhea (Gastrointestinal disorders) | 14
Dizziness (Nervous system disorders) | 18
Dry eye (Eye disorders) | 4
Dry mouth (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Dysgeusia (Nervous system disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Ear pain (Ear and labyrinth disorders) | 2
Edema limbs (General disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Eye pain (Eye disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 31
Fever (General disorders) | 10
Flatulence (Gastrointestinal disorders) | 1
Generalized weakness (Musculoskeletal and connective tissue disorders) | 16
Headache (Nervous system disorders) | 10
Hearing impaired (Ear and labyrinth disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypotension (Vascular disorders) | 1
Insomnia (Psychiatric disorders) | 11
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 15
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Nausea (Gastrointestinal disorders) | 29
Neutrophil count decreased (Investigations) | 10
Non-cardiac chest pain (General disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 2
Pain (General disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20
Papulopustular rash (Infections and infestations) | 1
Paresthesia (Nervous system disorders) | 20
Pelvic pain (Reproductive system and breast disorders) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 3
Platelet count decreased (Investigations) | 4
Proctitis (Gastrointestinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Rash pustular (Skin and subcutaneous tissue disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 9
Rectal pain (Gastrointestinal disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Thromboembolic event (Vascular disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 1
Tremor (Nervous system disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 6
Urinary tract pain (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 5
Vaginal hemorrhage (Reproductive system and breast disorders) | 7
Vaginal pain (Reproductive system and breast disorders) | 3
Vascular access complication (Injury, poisoning and procedural complications) | 1
Vomiting (Gastrointestinal disorders) | 20
Watering eyes (Eye disorders) | 1
Weight loss (Investigations) | 12
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
White blood cell decreased (Investigations) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT01676818/Prot_SAP_000.pdf